CLINICAL TRIAL: NCT02021669
Title: Omega-3 for Depression and Other Cardiac Risk Factors-2
Brief Title: Omega-3 for Depression and Other Cardiac Risk Factors - 2
Acronym: Omega-3(2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201309002; R01HL117805 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: Antidepressive agents; Coronary disease; Depression; Depressive disorder; Fatty Acids, Omega-3
MeSH Terms: conditions — Depression; Coronary Disease; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 supplement (Experimental): Two grams of the EPA form of omega-3 plus 50 mg of sertraline daily for 10 weeks
  Interventions: Drug: Omega-3 supplement
- Placebo (Placebo Comparator): Two grams of corn oil plus 50 mg of sertraline daily for 10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 supplement — Two grams of the EPA form of omega-3 daily and 50 mgs of sertraline daily for 10 weeks
  Other Names: EPA Plus Minami Nutrition
  Arms: Omega-3 supplement
Drug: Placebo — Two grams of corn oil plus 50 mg of sertraline daily for 10 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this 10 week randomized, placebo-controlled, double-blind clinical trial is to determine whether antidepressant augmentation with two grams of EPA omega-3 per day is superior to antidepressant therapy alone for major depression in patients with coronary heart disease (CHD).

DETAILED DESCRIPTION:
Depression increases the risk for cardiac morbidity and mortality 2-4 fold in patients with coronary heart disease (CHD). Recent clinical trials have tested standard treatments for comorbid depression in patients with CHD, and some have evaluated their effects on cardiac morbidity and mortality. Most of these trials have shown that standard treatments have only modest effects on depression and have produced relatively small differences between the intervention and control condition. Consequently, they have been unable to determine whether effective treatment of depression can improve cardiac outcomes. Low dietary intake and low plasma phospholipid or erythrocyte levels of two omega-3 fatty acids(FAs), eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), are associated with depression and other cardiac risk markers. There is growing evidence from small psychiatric trials that the efficacy of standard antidepressants can be improved by coadministration of an omega-3 FA formulation containing at least 1 gram of EPA. The purpose of the proposed research is to determine whether antidepressant augmentation with this omega-3 formulation is superior to antidepressant therapy alone for major depression in patients with CHD. The proposed study is a randomized, placebo-controlled, double-blind clinical trial. Consenting patients with established coronary heart disease who meet the Diagnostic Statistical Manual (DSM)-5 criteria for a major depressive episode will undergo a baseline evaluation and then be randomly assigned to receive either 50 mg/day of sertraline plus omega-3 FA or 50 mg/day of sertraline plus placebo for 10 weeks. At baseline and after 10 weeks, participants will complete assessments of depression, 24 hour ambulatory ECG monitoring to measure 24 hour heart rate and heart rate variability, and blood draws to measure procoagulant and proinflammatory markers and blood levels of EPA, DHA, other omega-3 FAs, and the omega-6 FAs. If sertraline plus this omega-3 formulation significantly reduces depression compared to sertraline plus placebo, and if it improves or at least does not worsen other cardiovascular risk markers, this study will provide a strong basis for proposing a multicenter clinical trial of sertraline augmented with omega-3 to determine whether treatment of depression can improve survival in patients with CHD and depression.

ELIGIBILITY:
Inclusion Criteria:

* Documented coronary heart disease
* Diagnosis of major depression based on structured interview

Exclusion Criteria:

* Moderate to severe cognitive impairment
* Meets DSM-5 criteria for depressive disorder due to a general medical condition or medication
* Major Axis I psychiatric disorder other than unipolar depression or an anxiety disorder, a high risk of suicide, or current substance abuse other than tobacco;
* Not expected to survive one year or physically unable to tolerate the study protocol
* Known sensitivity to sertraline or omega-3, or an allergy to fish oil or shellfish
* Taking an antidepressant or an omega-3 supplement at baseline
* Exempted by their cardiologist or primary care physician
* Refuses to provide informed consent
* Participating in a competing protocol or trial

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Carney, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carney RM, Freedland KE, Rubin EH, Rich MW, Steinmeyer BC, Harris WS. A Randomized Placebo-Controlled Trial of Omega-3 and Sertraline in Depressed Patients With or at Risk for Coronary Heart Disease. J Clin Psychiatry. 2019 Jun 4;80(4):19m12742. doi: 10.4088/JCP.19m12742. PMID 31163106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega-3 Supplement | Placebo
Started | 71 | 73
Completed | 64 | 70
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Supplement | Placebo | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 46 | 95
  >=65 years | 22 | 27 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.6) | 60.5 (9.3) | 59.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 45 | 43 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 27 | 48
  White | 44 | 45 | 89
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 71 | 73 | 144

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item self-report inventory of depression symptoms. The minimum and maximum values for the BDI-II are (0-63). For both instruments, the higher the scores, the greater the severity of depression.
Time Frame: Change from baseline to 10 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 Supplement | Placebo
Number analyzed (Participants) | 71 | 73
score on a scale
  Baseline | 29.9 (9.0) | 29.1 (8.8)
  Post Treatment (10 Weeks) | 11.0 (9.9) | 9.1 (7.7)

2. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D, 17)
Description: The HAM-D, 17 is a 17-item, observer-rated measure of depression symptoms. The minimum and maximum values for the HAM-D, (0-52). For both instruments, the higher the scores, the greater the severity of depression.
Time Frame: Change from baseline to 10 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 Supplement | Placebo
Number analyzed (Participants) | 71 | 73
score on a scale
  Baseline | 17.4 (5.4) | 17.0 (5.0)
  Post Treatment (10 Weeks) | 7.1 (7.0) | 6.2 (5.5)

ADVERSE EVENTS:
Time Frame: Each participant was followed for fourteen weeks (ten weeks of treatment plus a final call 4 weeks after the end of treatment)
Arm/Group | Omega-3 Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 35/71 | 32/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Supplement (N=71) | Placebo (N=73)
Nausea (General disorders) | 15 (15) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 15 (15)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Increased flatulence (Gastrointestinal disorders) | 2 (2) | 3 (3)
Increased sleepiness (General disorders) | 8 (8) | 5 (5)
Fatigue (General disorders) | 4 (4) | 3 (3)
Dizziness (General disorders) | 3 (3) | 2 (2)
Insomnia (General disorders) | 2 (2) | 0 (0)
Hand Tremors (Nervous system disorders) | 2 (2) | 3 (3)
Decreased sexual interest/performance (General disorders) | 1 (1) | 2 (2)
Less emotionally responsive (Social circumstances) | 3 (3) | 2 (2)
Headaches (General disorders) | 3 (3) | 6 (6)
Increased anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1)
Increased sweating (General disorders) | 2 (2) | 3 (3)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bad taste in mouth (General disorders) | 1 (1) | 3 (3)
Burping (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02021669/Prot_SAP_ICF_000.pdf